CLINICAL TRIAL: NCT01913366
Title: Case Management and Problem Solving Therapy for Depressed Older Adults
Brief Title: Senior Peer Alliance for Rural Research On Wellness
Acronym: SPARROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AG043584-01A1 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: MDD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CM-PST (Experimental): If you are assigned to CM-PST, you will be working with the same care manager from your introductory session. The care manager will continue to work with you on your problem-solving plan. Additionally, you will receive case management services.
  Interventions: Behavioral: CM-PST
- SG-PST (Experimental): If you are assigned to SG-PST, you will continue to work on your problem-solving plan, using the self-guided materials provided to you during the introductory session. Additionally, you will be partnered with a senior peer counselor who will support you in your SG-PST efforts.
  Interventions: Behavioral: SG-PST

INTERVENTIONS:
Behavioral: CM-PST
  Arms: CM-PST
Behavioral: SG-PST
  Arms: SG-PST

SUMMARY:
Dr. Brooke Hollister, Ph.D. from the department of Social and Behavioral Sciences at the University of California, San Francisco is conducting a study comparing two types of interventions for treating depression in rural older adults.

DETAILED DESCRIPTION:
If you are eligible to participate in the study after completing the screening assessment, and if you choose to continue on, we will randomize you (like a flip of a coin) to receive either 12 weeks of case management combined with problem solving therapy (CM-PST) with a social worker or 12 weeks of self-guided problem solving therapy (SG-PST) with support from a senior peer counselor.

As part of your participation in the study you will participate in three 1.5 hour assessment interviews of psychological and neuropsychological functioning (similar to your screening assessment) prior to your first week of treatment (baseline), two weeks after your final session (week 14), and three months after your final session (week 24). Additionally, you will participate in three shorter assessment interviews of psychological functioning, which will be conducted at weeks 3 and 6. These assessments will take approximately 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Residence in rural Tuolumne, Calaveras, San Joaquin or Stanislaus Counties;
* Diagnosis: Major depression, unipolar (by SCID ascertained DSM-IV criteria);
* Severity of depression: A PHQ-9>10 or a 24-Item HDRS>19;
* Need for social services: CANE score> 2, i.e. at least one unmet need;

Exclusion Criteria:

* Psychotic depression by SCID-IV, i.e., presence of delusions;
* High suicide risk, i.e. intent or plan to attempt suicide in near future;
* Presence of any Axis I psychiatric disorder or substance abuse other than unipolar major depression;
* Axis II diagnosis of antisocial personality (by SCID-P and DSM-IV);
* History of psychiatric disorders other than unipolar major depression or generalized anxiety disorder (including bipolar disorder, hypomania, and dysthymia);
* Dementia: MMSE below 24 or clinical diagnosis of dementia by DSM-IV;
* Acute/severe medical illness (delirium, metastatic cancer, de-compensated cardiac, liver or kidney failure, stroke or myocardial infarction) 3 months prior to entry; or use of drugs causing depression, (steroids, reserpine, alphamethyl-dopa, tamoxiphen, vincristine);
* Inability to perform any of the ADLs (MAI: ADL subscale) even with assistance (walking with a cane is not an exclusion criterion)
* Inability to speak English;
* Aphasia interfering with communication;

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD) | Baseline
  A multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.
Hamilton Rating Scale for Depression (HRSD) | Week 3
  A multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.
Hamilton Rating Scale for Depression (HRSD) | Week 6
  A multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.
Hamilton Rating Scale for Depression (HRSD) | Week 12
  A multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.
WHO Disability Assessment Schedule 2.0 (WHODAS-II) | Week 0
  Generic assessment instrument for health and disability
WHO Disability Assessment Schedule 2.0 (WHODAS-II) | Week 3
  Generic assessment instrument for health and disability
WHO Disability Assessment Schedule 2.0 (WHODAS-II) | Week 6
  Generic assessment instrument for health and disability
WHO Disability Assessment Schedule 2.0 (WHODAS-II) | Week 12
  Generic assessment instrument for health and disability

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Hollister, Ph.D., Principal Investigator — University of California, San Francisco; Patricia Arean, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Catholic Charities Motherlode Office- Sonora, Sonora, California, United States